CLINICAL TRIAL: NCT07086586
Title: Relationship Between Isokinetic Hip Muscles Performance Parameters and Balance in Patients With Chronic Ankle Instability
Status: Completed | Type: Observational
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Gehad Mohamed Mahmoud Mubarak, Bsc. of physiotherapy, General Committee of Teaching Hospitals and Institutes, Egypt
Other Study IDs: Cairo university 1
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2023-07

CONDITIONS: Chronic Ankle Instability, CAI
Keywords: SEBT , balance, eccentric hip contraction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- one shot study: isokinetic eccentric muscle assessment and star excursion balance test

SUMMARY:
Observational, Cross- sectional study (one shot study), design will used (Correlation study) This study aims to investigate the relationship between hip muscles performance and balance in patients with chronic ankle instability using the Star Excursion Balance Test (SEBT) and Isokinetic biodex system III.

this study is to answer the question ; Is there a relationship between hip muscles (extensors/flexors, abductors /adductors, internal rotator/ lateral rotator) performance and balance in patients with chronic ankle instability?

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18 and 40 years from both genders.
2. Had a history of at least one significant lateral ankle sprain to the same side that resulted in pain and loss of function of more than one day.
3. Had a history of at least two episodes of 'giving way' in the past six months.
4. Each member of the CAI group will require to answer yes to at least 5 questions on the Ankle Instability Instrument (AII) questionnaire and score 24 on the Cumberland Ankle Instability Tool (CAIT)

Exclusion Criteria:

1. A history of neural or vestibular disorders.
2. Previous lower limb surgeries
3. Trauma to the lower limbs for at least 3 months prior to the study;
4. Physiotherapy within the last 3 months or current participation in supervised physical rehabilitation.
5. Consumed drugs or alcohol within 24 hours prior to testing that could interfere with performance.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited in the study from outpatient clinic of Cairo University and orthopedic physician.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2024-10-19 (Actual)

PRIMARY OUTCOMES:
hip muscle performance | one time
  flexion, extension, abduction , adduction , external rotation ,internal rotation

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided